CLINICAL TRIAL: NCT06546891
Title: Using an Adaptive Rower for People Using Motorized Wheelchairs to Improve Cardiovascular Fitness
Brief Title: Using an Adaptive Rower for People Using Motorized Wheelchairs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Foundation for Physical Therapy, Inc. (Industry)
Responsible Party: Principal Investigator, Elizabeth Regan, Clinical Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00137469
Record Dates: First submitted 2024-08-02; First posted 2024-08-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: People Who Use Motorized Wheelchairs for Mobility
Keywords: motorized wheelchair; exercise; adaptive fitness; rowing
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Single Group Case Series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Intervention Arm - Adaptive Rowing (Experimental): 12 supervised and coached sessions of 10-20 minutes of moderate to vigorous exercise using an adaptive rower.
  Interventions: Behavioral: Adaptive Rowing

INTERVENTIONS:
Behavioral: Adaptive Rowing — 12 supervised and coached sessions of 10-20 minutes of moderate to vigorous exercise using an adaptive rower.

SUMMARY:
The goal of this clinical trial are to determine the feasibility and impact of an adaptive rower exercise intervention for adults who use motorized wheelchairs for mobility.

The main question[s] it aims to answer are:

1. What is the impact on participant's cardiovascular endurance, and perception of mobility and quality of life?
2. Is the intervention feasible, acceptable and safe?

examine feasibility of the adaptive rower intervention through measures of acceptability, adherence, intensity and safety for adults who use motorized wheelchairs for mobility.

Participants will complete 12 sessions of 10-20 minutes of supervised and coached moderate to vigorous activity using the adaptive rower over a seven week period. Participants will complete pre- and post- outcome assessments of cardiovascular fitness, and outcome surveys,

DETAILED DESCRIPTION:
A rolling prospective clinical trial with a target population of 10 participants in the Columbia, South Carolina area will evaluate the impact of the adaptive rower on cardiovascular fitness, participant perception and feasibility for people who use motorized wheelchairs.

Participants will be screened for inclusion/exclusion criteria, perform initial outcome measures and instructions on rowing in the first visit, and then have 12 exercise sessions over 6 or 7 weeks, followed by a final visit for final outcome measures. All research will occur at the University of South Carolina Rehab Lab in the public health research center building.

Over the 6-7 week intervention period, participants will exercise approximately two times per week, with two additional visits available in week 7 for any missed sessions to fulfill the 12-visit dosage. Session data will include measures of heart rate, 0-10 Borg rate of perceived exertion (RPE), and power output (rower output in watts). The session goal is to maintain moderate-vigorous intensities (5-8 on the Borg RPE scale) with individually modifiable intervals of work and rest with the goal of 10-20 minutes of moderate-vigorous physical activity total per session depending on the individual's initial fitness levels (as judged by self-reported activity level and performance on the initial six-minute arm test) and progressed as able. After completing the intervention period, participants will return for final evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Use a motorized wheelchair for mobility
* Able to perform a rowing motion with upper extremities with or without grip aids

Exclusion Criteria:

* Existing pressure sores
* Increasing pain with rowing motion
* Unstable angina
* Uncontrolled arrythmia
* Acute illness with fever
* Blood pressure above 180/100 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Six Minute Arm Test | Study Start (Week 1) and at Study Completion (week 7-8)
  Submaximal fitness test using an upper body ergometer. Maximum power, maximum rate of perceived exertion and maximum heart rate are recorded. Higher power, lower RPE and lower maximum heart rate is better outcome
Spinal Cord Injury Functional Inventory basic mobility, motorized wheelchair mobility and resilience subscales | Study Start (Week 1) and at Study Completion (week 7-8)
  Scores from 0-100% where mean scores for population is 50%, higher score better outcome

SECONDARY OUTCOMES:
System Usability Scale | Study Completion (week 7-8)
  a standardized 10-question survey for perception of usability, scored from 0-100%, higher score, better outcome
Physical Activity Enjoyment Scale-Short (PACES-S) | Study Completion (week 7-8)
  a standardized 4-question survey for perception of enjoyment of a physical activity intervention, scale is 1 (strongly disagree) to 5 (strongly agree), total score 4-20 with higher score as better outcome
Heart Rate (beats per minute), mean and range at rest, mean and range during rowing | 2 x a week through study completion, 7-8 weeks
  Heart rate will be recorded at rest and throughout the exercise intervention using a polar heart rate monitor and actigraph. Heart rate near target zone, better outcome
Rate of Perceived Exertion (RPE)-Borg 6-20 Scale | 2 x a week through study completion, 7-8 weeks
  RPE will be verbally stated by participant and recorded by study personnel at beginning, mid and end of steady state portion, and at each interval for interval exercise. (RPE, 6-20, higher means higher intensity) RPE within target zone of moderate intensity (12-14) better outcome
Pain Scale (0-10 visual analog scale) and body location of pain verbalized by participant and recorded by study personnel | 2 x a week through study completion, 7-8 weeks
  participant complaints of discomfort or pain verbally stated along with location. Higher means worse pain, lower is better outcome

OTHER OUTCOMES:
Short Self-Efficacy for Exercise Scale | Study Start (Week 1) and at Study Completion (week 7-8)
  A standardized 9-question survey to measure participant confidence in being able to exercise under a variety of conditions. Scores are 0-90 where higher scores indicate better outcome .

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Public Health Research Center, Columbia, South Carolina
  - Still Hopes Retirement Community, West Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be part of dissemination of project results and be shared on open science framework. Data shared would be basic demographics (age, sex), pre and post outcome measures (six minute arm test time, spinal cord functional index score, PROMIS Scales for wheelchair mobility and resilience), session data (minutes of rowing, minutes of rest time, RPE ratings, heart rate data, pain/soreness ratings)
Time Frame: Data will be available after completion of the study when dissemination occurs; and will be available indefinitely
Access Criteria: website
URL: http://osf.io/

DOCUMENTS (1):
  • Informed Consent Form (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT06546891/ICF_000.pdf